CLINICAL TRIAL: NCT00633646
Title: Effect of Protein-Restricted Diet on Nitrogen Balance and Residual Renal Function in PD Patients
Brief Title: Effect of Protein-Restricted Diet on Nitrogen Balance and Residual Renal Function in Peritoneal Dialysis (PD) Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Qiang Yao, Renji Hospital, Shanghai Jiaotong University, School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05PJ14057(Shanghai, China)
Record Dates: First submitted 2008-02-22; First posted 2008-03-12 (Estimated); Last update posted 2008-04-28 (Estimated); Status verified 2008-03

CONDITIONS: Chronic Kidney Disease; Peritoneal Dialysis
Keywords: nitrogen balance; malnutrition; chronic kidney disease; diet; glomerular filtration rate
MeSH Terms: conditions — Renal Insufficiency, Chronic; Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): low protein diet
  Interventions: Dietary Supplement: diets contained different levels of protein
- 2 (Active Comparator): low protein diet with keto acids
  Interventions: Dietary Supplement: diets contained different levels of protein
- 3 (Active Comparator): high protein diet
  Interventions: Dietary Supplement: diets contained different levels of protein

INTERVENTIONS:
Dietary Supplement: diets contained different levels of protein — diets contain protein in the range of 0.6-0.8 or 1.0-1.2 g/kg/d
  Other Names: LP; sLP; HP

SUMMARY:
Current therapy recommendations suggest a low protein diet to preserve residual renal function (RRF) before the start of dialysis, but a higher protein intake during dialysis to prevent protein-energy wasting (PEW). We conducted a randomized trial to test whether low protein intake also during treatment with peritoneal dialysis (PD) would be safe and associated with a preserved RRF.

DETAILED DESCRIPTION:
Dietary protein is the major source of nitrogen excreted as urea by the kidney, and a decreased protein intake has been associated with a retardation of kidney function loss in non-dialysis chronic kidney disease (CKD) patients. While a low protein diet is recommended to end-stage renal disease (ESRD) patients before the start of dialysis to preserve residual renal function(RRF), current therapy recommendations in dialysis are for a normal protein intake of no less than 1.2 g of protein/kg ideal body weight (IBW)/day to prevent protein-energy wasting (PEW).

We hypothesized that a lower protein intake would be safe and able to slow the loss of RRF also in dialysis patients and conducted two prospective, randomized trials involving a total of 94 peritoneal dialysis (PD) patients to test our hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* age 18-80 years
* stable peritoneal dialysis since at least 1 month
* with renal function

Exclusion Criteria:

* a high probability (assessed by the recruiting physician) of receiving a kidney transplant within one year
* overt infection within the last month
* poor compliance in previous dietary prescriptions or irregular check-ups
* persistent anorexia, vomiting or diarrhea within the last month
* a CRP of more than 30 mg/dL
* presence of wasting diseases such as cancer or tuberculosis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2006-01; Primary Completion 2008-01 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
nitrogen balance,residual renal function and nutritional status | 10 day and 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Yao Qiang, MD, Ph.D, Principal Investigator — RenJi Hospital